CLINICAL TRIAL: NCT01808053
Title: Assessment of the BodyGuardian Remote Monitoring Platform in Elderly Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH); Preventice (Industry)
Responsible Party: Principal Investigator, Charles J. Bruce, Principal Investigator, Mayo Clinic
Other Study IDs: 12-008639; R01AG041676 (NIH)
Record Dates: First submitted 2013-03-07; First posted 2013-03-08 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy older and independently living adults: The BodyGuardian remote health monitoring system will used by healthy older and independently living adults
  Interventions: Device: BodyGuardian remote health monitoring system

INTERVENTIONS:
Device: BodyGuardian remote health monitoring system — The remote health management system connects personal health sensors with secure mobile communication devices. It is also able to give immediate feedback to the user. The solution is a multi-tiered mobile health platform. The front-end includes an adhesive snap-strip body sensor (BodyGuardian) that can measure HR, ECG, respiration rate (RR), and activity which is FDA approved for detection of non-lethal cardiac arrhythmias. It can wirelessly communicate with off-body sensors such as a BP cuff and scale to incorporate BP and weight data based on automated algorithms and can solicit symptoms from the user. It can also be used as an event recorder inputting symptoms and recording simultaneous physiologic data.

SUMMARY:
To adapt and refine the BodyGuardian remote health monitoring system to acquire ECG, Heart rate (HR), activity and breathing data, which will be integrated with weight, blood pressure and symptom data, in subjects in an independent living center, with wireless transmission of data to a central data analysis hub.

DETAILED DESCRIPTION:
The elderly are facing an increasing prevalence of chronic disease and rapidly escalating healthcare costs threatening independent living. Congestive heart failure (CHF) is a growing health epidemic and is associated with significant morbidity, mortality and cost. Mayo Clinic and Preventice have developed a non-invasive, minimally obtrusive, interactive remote monitoring platform. It enables on-body monitoring and integration of ECG, heart rate, breathing, and activity, with measures of weight and blood pressure. It is designed as a platform for physician directed patient self-management. This technology may be useful in monitoring CHF patients. Our overall objective is to adapt, refine, test and validate this technology in subjects in an independent living center, with wireless transmission of data to a central data analysis hub.

ELIGIBILITY:
Inclusion Criteria:

* Resident at independent living facility
* Adequate phone service
* Healthy with life anticipated survival >than one year

Exclusion Criteria:

* Skin reaction/allergies to adhesives
* Have implantable pacemaker and/or defibrillator or have a bed partner with an implantable pacemaker

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy older adults living at an independent living center.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with successful data transfer at the end of 30 day monitoring period. | approximately at the end of 30 day monitoring period
  Data collected will be reviewed by engineering collaborators.

CONTACTS AND LOCATIONS:
Overall Officials: Charles J Bruce, MBChB, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States